CLINICAL TRIAL: NCT05686668
Title: Evolution of the Sensory Profile in Depression
Acronym: DEPSENS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Aude Paquet, Principal Investigator, Psychomotor Therapist, Centre Hospitalier Esquirol
Other Study IDs: CHEsquirol
Record Dates: First submitted 2022-12-15; First posted 2023-01-17 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Adolescent Adult Sensory Profile; Sensory Profiles; Coping
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AASP
  Interventions: Other: assessment by scales

INTERVENTIONS:
Other: assessment by scales — Assessment from many scales: AASP, HARS, HDRS, CORE, EES, CISS, SHAPS at V1 Assessment from many scales: AASP, HARS, HDRS, CORE, EES, SHAPS at V2

SUMMARY:
The perception of the environment through the study of sensory awareness is important to understand the adaptive or symptomatological behaviors (e.g., withdrawal, increased activity level, stimulation seeking, etc.). Sensory processing disorders, such as hypersensitivities or hyposensitivities, have been described in people with depression using the Adolescent Adult Sensory Profile scale. In a recent study, similar results consistent with extreme sensory profiles (hypersensitivity, hyposensitivity, sensation avoidance) in adults with a major depressive disorder were observed. The evolution over time of the sensory profile in people with a depressive disorder is not known. It is currently unknown whether these extreme sensory processing profiles are stable over time or whether they may evolve with the depressive symptomatology to normalize with clinical improvement.

This knowledge could have an important impact both on the symptomatological expression of the disorder, its recognition, and also on the management of the patient. The investigators aim to study the evolution over time of the sensory profile of depressed subjects hospitalized using the ASSP. The behavioral responses of individuals with sensory processing disorder may be related to the coping strategies of these individuals with their living environment. In a second step, the investigators will study the second step the sensory profile of subjects with depression according to their coping strategies, their living environment and their clinical characteristics (anxiety (anxiety, psychomotor slowing, self-esteem, anhedonia).

DETAILED DESCRIPTION:
Main objective To compare the sensory profiles, i.e., the distribution of sensory processing patterns at each quadrant of the AASP, of subjects with major depressive disorder at the beginning of hospitalization (V1), and 3 months later (V2).

Secondary objectives

* Objective 1: To describe at V1 and V2, the sensory profiles according to the clinical characteristics (anxiety, depression, psychomotor slowing, self-esteem, anhedonia); a difference in the relationship between the clinical scales and the quadrants (AASP) at V2 and V1 could be observed.
* Objective 2: To look for a difference in sensory profile at V2 according to clinical improvement
* Objective 3: To compare, at V1, the distribution of processing patterns of sensory profiles for each quadrant of the AASP, according to coping styles (CISS).
* Objective 4: To compare the distribution of processing patterns of sensory profiles sensory profiles for each quadrant of the AASP, according to socio-demographic characteristics: gender, age group, professional category, type of type of housing, environment, family situation
* Objective 5: To look for a difference in the distribution of the processing patterns sensory profiles between the first inclusion visit (V1) and 3 months (V2), according to the type of drug treatment (molecules and classes) and non (psychotherapy, relaxation, rTMS, ECT) Inclusion criteria
* Male or female, 18 to 65 years of age
* who have given informed consent
* with a diagnosis of a major depressive disorder according to the DSM-5 criteria
* in full hospitalization for less than 10 days in the care units of the Esquirol Hospital

Non inclusion criteria

* Psychiatric comorbidity (personality disorder, addiction other than tobacco, eating disorder, bipolar disorder, obsessive-compulsive disorder, schizophrenia and related disorders)
* Sensory or neurological disability
* Inability to understand the questionnaires and information related to the study
* Hospitalization under constraint, pregnancy, subjects under guardianship or curatorship, lack of social protection

Outcome Measures Primary endpoints

- AASP at V1 and V2 Secondary endpoints

1. AASP, HARS, HAM-D, CORE, EES-10, SHAPS at V1 and V2
2. AASP, HAM-D at V2
3. AASP, ISSC
4. AASP scores and socio-demographic characteristics (age, sex ratio, living environment, family status, housing)
5. AASP scores and treatments at V1 and V2

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age
* who have given informed consent
* with a diagnosis of a major depressive disorder according to the DSM-5 criteria
* in full hospitalization for less than 10 days in the care units of the Esquirol Hospital

Exclusion Criteria:

* Psychiatric comorbidity (personality disorder, addiction other than tobacco, eating disorder, bipolar disorder, obsessive-compulsive disorder, schizophrenia and related disorders)
* Proven sensory or neurological disability
* Inability to understand the questionnaires and information related to the study
* Hospitalization under constraint, pregnancy, subjects under guardianship or curatorship, lack of social protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized poeple for a major depressive disorder
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Adolescent Adult Sensory Profile score | day 0 and 3 months
  measure a change in Adolescent Adult Sensory Profile score between he beginning of hospitalization and 3 months

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale score | day 0 and 3 months
  measure a change in Adolescent Adult Sensory Profile score according to the HARS
number of participants with psychomotor retardation | day 0 and 3 months
  measure a change in Adolescent Adult Sensory Profile score according to the psychomotor retardation-CORE scale
Snaith-Hamilton pleasure scale score | day 0 and 3 months
  measure a change in Adolescent Adult Sensory Profile score according to SHAPS score
Coping Inventory for Stressful Situations score | day 0
  the distribution of processing patterns of sensory profiles were compared according to coping styles based on CISS score
number of participants living in country | day 0
  compare the Adolescent Adult Sensory Profile score according to living environment (country or town)
number of participants living lonely | day 0
  compare the Adolescent Adult Sensory Profile score according to the family status (living alone or with people)
Treatments | day 0 and 3 months
  measure a change in Adolescent Adult Sensory Profile score according to the traitments (antidepressant, anxiolytic, neuroleptic, psycho-corporal therapy)

CONTACTS AND LOCATIONS:
Locations (1):
- CH Esquirol, Limoges, France

IPD SHARING:
Plan to Share IPD: No